CLINICAL TRIAL: NCT01981551
Title: Phase II Trial of the Gamma-Secretase Inhibitor PF-03084014 in Adults With Desmoid Tumors/Aggressive Fibromatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alice Chen, M.D., Associate Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140007; 14-C-0007
Record Dates: First submitted 2013-10-31; First posted 2013-11-11 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Desmoid Tumors; Aggressive Fibromatosis
Keywords: Desmoid Tumor; Aggressive Fibromatosis; Gamma-secretase Inhibitor; Notch Pathway
MeSH Terms: conditions — Desmoid Tumors | interventions — nirogacestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-03084014 in Desmoid Tumors/Aggressive Fibromatosis (Experimental): PF-03084014 will be administered orally at 150 mg twice a day in 21-day cycles
  Interventions: Drug: PF-03084014

INTERVENTIONS:
Drug: PF-03084014 — Treatment with the selective small-molecule >=-secretase inhibitor PF- 3084014 caused significant tumor shrinkage in patients with unresectable desmoid tumors in an early-phase clinical trial.

SUMMARY:
Background:

* Desmoid tumors (also known as aggressive fibromatosis), are rare, locally invasive, slow-growing soft-tissue tumors. The disease can be either asymptomatic or be associated with severe loss of organ function and significant morbidity.
* Treatment with the selective small-molecule Gamma-secretase inhibitor PF-03084014 caused significant tumor shrinkage in patients with unresectable desmoid tumors in an early phase clinical trial.
* The Notch pathway is a key regulator of cell differentiation, proliferation and apoptosis; aberrant signaling via the Notch pathway is associated with carcinogenesis.

Objectives:

* Primary: Determine the response rate (Complete Response (CR)+Partial Response (PR)) of PF-03084014 in patients with desmoid tumors/aggressive fibromatosis
* Secondary: Assess symptom measures at baseline and on study; perform genotyping for germline and somatic mutations in adenomatous polyposis coli gene (APC) and catenin-beta 1 (CTNNB1) genes; correlate clinical response to therapy with genotyping data; and assess modulation of the Notch pathway by evaluating notch response genes in tumor biopsies at baseline and after drug administration

Eligibility:

* Age greater than or equal to18; histologically confirmed desmoid tumor not amenable to curative resection or definitive radiation therapy that has progressed after receiving at least one line of standard treatment; adequate organ function
* Willingness to provide blood samples and 10 unstained slides or a tumor block for genetic research studies

Study Design:

* This is an open-label Phase II trial of PF-03084014; study drug will be administered orally at 150 mg twice a day in 21-day cycles
* Optional tumor biopsies for research purposes will be performed at baseline prior to study treatment and at the beginning of cycle 7 (+/- one cycle)
* Restaging scans (magnetic resonance imaging (MRI) with diffusion weighting) will be performed at baseline, at the end of cycles 1 and 6, and then every 6 cycles
* Health-related quality of life (HRQOL)/symptom questionnaires will be administered at baseline and at each Clinical Center visit

DETAILED DESCRIPTION:
Background:

* Desmoid tumors (also known as aggressive fibromatosis), are rare, locally invasive, slow-growing soft-tissue tumors. The disease can be either asymptomatic or be associated with severe loss of organ function and significant morbidity.
* Treatment with the selective small-molecule Gamma-secretase inhibitor PF-03084014 caused significant tumor shrinkage in patients with unresectable desmoid tumors in an early phase clinical trial.
* The Notch pathway is a key regulator of cell differentiation, proliferation and apoptosis; aberrant signaling via the Notch pathway is associated with carcinogenesis.

Objectives:

* Primary: Determine the response rate (Complete Response (CR)+Partial Response (PR)) of PF-03084014 in patients with desmoid tumors/aggressive fibromatosis
* Exploratory: Assess symptom measures at baseline and on study; perform genotyping for germline and somatic mutations in adenomatous polyposis coli gene (APC) and catenin-beta 1 (CTNNB1) genes; correlate clinical response to therapy with genotyping data; and assess modulation of the Notch pathway by evaluating notch response genes in tumor biopsies at baseline and after drug administration

Eligibility:

* Age greater than or equal to18; histologically confirmed desmoid tumor not amenable to curative resection or definitive radiation therapy that has progressed after receiving at least one line of standard treatment; adequate organ function
* Willingness to provide blood samples and 10 unstained slides or a tumor block for genetic research studies

Study Design:

* This is an open-label Phase II trial of PF-03084014; study drug will be administered orally at 150 mg twice a day in 21-day cycles
* Optional tumor biopsies for research purposes will be performed at baseline prior to study treatment and at the beginning of cycle 7 (+/- one cycle)
* Restaging scans (computed tomography (CT) scan of the known site of disease) will be performed at baseline and then every 6 cycles (+/- one cycle)
* Optional magnetic resonance imaging (MRI) scans may be performed prior to start of study treatment, end of cycle 1, and every 6 cycles (at the same times as the CT scans)
* Health-related quality of life (HRQOL)/symptom questionnaires will be administered at baseline and at restaging

ELIGIBILITY:
* INCLUSION CRITERIA:

2.1.1.1 Patients must have histologically confirmed desmoid tumor confirmed by the Laboratory of Pathology, National Cancer Institute (NCI), that has progressed after receiving at least one line of standard treatment and that is not amenable to surgical resection or definitive radiation therapy.

2.1.1.2 Willingness to provide blood samples and 10 unstained slides or a tumor block for genetic research studies.

2.1.1.3 Any line of therapy with prior desmoid therapy, including radiotherapy, should have been completed at least 2 weeks before study entry and all toxicities must have resolved at least to eligibility levels.

2.1.1.4 Age greater than or equal 18 years; because no dosing or adverse event data are currently available on the use of PF-03084014 in patients <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials.

2.1.1.5 Eastern Cooperative Oncology Group (ECOG) performance status less than or equal 2.

2.1.1.6 Life expectancy > 3 months.

2.1.1.7 Patients must have normal organ and marrow function as defined below:

* -absolute neutrophil count greater than or equal 1,500/mcL
* -platelets greater than or equal 100,000/mcL
* -total bilirubin less than or equal 1.5 times institutional upper limit of normal
* -Aspartate aminotransferase (AST) Serum Glutamic Oxaloacetic Transaminase (SGOT)/Alanine aminotransferase (ALT) Serum glutamic-pyruvic transaminase (SGPT) less than or equal 5 times institutional upper limit of normal
* -creatinine < 1.5 times institutional upper limit of normal

OR

* -creatinine clearance greater than or equal 60 mL/min/1.73 m(2) for patients with creatinine levels >1.5 mg/dL
* -hemoglobin greater than or equal 9 g/dL

2.1.1.8 Patients must be able to swallow whole tablets or capsules with no gastrointestinal (GI) condition affecting absorption; nasogastric or G-tube administration is not allowed.

2.1.1.9 The effects of PF-03084014 on the developing human fetus are unknown. For this reason and because >=-secretase inhibitors are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation and for at least 6 months after dosing with study drugs ceases. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception for the duration of study participation, and 6 months after completion of study drug administration.

2.1.1.10 Ability to understand and the willingness to sign a written informed consent document.

2.1.1.11 Evidence of measurable disease by computed tomography (CT) scan. Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than or equal 20 mm by chest x-ray, as greater than or equal 10 mm with CT scan, or greater than or equal 10 mm with calipers by clinical exam.

EXCLUSION CRITERIA:

2.1.2.1 Patients who are receiving any other investigational agents. Concurrent mediations that the patient is taking will be reviewed by the principal investigator (PI) to assess safety and eligibility.

2.1.2.2 Prior treatment with Gamma-secretase inhibitors or anti-notch antibody therapy.

2.1.2.3 Uncontrolled intercurrent illness including, but not limited to, serious infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

2.1.2.4 Corrected QT interval (QTc) interval of >470 msec at study entry; congenital long QT syndrome.

2.1.2.5 Pregnant women are excluded from this study because PF-03084014 is a Gamma-secretase inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with PF-03084014, breastfeeding should be discontinued if the mother is treated with PF-03084014.

2.1.2.6 Patients with gastrointestinal conditions that might predispose for drug intolerability or poor drug absorption (e.g., inability to take oral medication or a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, malabsorption syndrome, and active peptic ulcer disease) are excluded. Subjects with ulcerative colitis, inflammatory bowel disease, or a partial or complete small bowel obstruction are also excluded, as are any patients who cannot swallow the tablet whole. Tablets must not be crushed or chewed; nasogastric or gastrostomy (G)-tube administration is not allowed.

2.1.2.7 Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with PF-03084014.

2.1.3 Recruitment Strategies

We have had multiple discussions with the Desmoid Tumor Research Foundation, Inc., who have various outreach efforts including patient meetings and webcasts. Senior executives of the Foundation have indicated strong interest in this trial and willingness to inform their members. We also have a network of referring physicians nationally that refers patients with solid tumors to our clinical program. Given our interest and trials for sarcomas, we have formed connections with centers that treat patients with mesenchymal malignancies. We will be informing all of these of the availability of this trial once it is open.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine H O'Sullivan Coyne, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Background] de Bree E, Keus R, Melissas J, Tsiftsis D, van Coevorden F. Desmoid tumors: need for an individualized approach. Expert Rev Anticancer Ther. 2009 Apr;9(4):525-35. doi: 10.1586/era.09.9. PMID 19374605
- [Background] Lev D, Kotilingam D, Wei C, Ballo MT, Zagars GK, Pisters PW, Lazar AA, Patel SR, Benjamin RS, Pollock RE. Optimizing treatment of desmoid tumors. J Clin Oncol. 2007 May 1;25(13):1785-91. doi: 10.1200/JCO.2006.10.5015. PMID 17470870
- [Background] Lewis JJ, Boland PJ, Leung DH, Woodruff JM, Brennan MF. The enigma of desmoid tumors. Ann Surg. 1999 Jun;229(6):866-72; discussion 872-3. doi: 10.1097/00000658-199906000-00014. PMID 10363901
- [Result] Kummar S, O'Sullivan Coyne G, Do KT, Turkbey B, Meltzer PS, Polley E, Choyke PL, Meehan R, Vilimas R, Horneffer Y, Juwara L, Lih A, Choudhary A, Mitchell SA, Helman LJ, Doroshow JH, Chen AP. Clinical Activity of the gamma-Secretase Inhibitor PF-03084014 in Adults With Desmoid Tumors (Aggressive Fibromatosis). J Clin Oncol. 2017 May 10;35(14):1561-1569. doi: 10.1200/JCO.2016.71.1994. Epub 2017 Mar 28. PMID 28350521
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0007.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PF-03084014 in Desmoid Tumors/Aggressive Fibromatosis
Started | 17
Completed | 8
Not Completed | 9
Not completed — Refused further treatment | 8
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | PF-03084014 in Desmoid Tumors/Aggressive Fibromatosis
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.02 (14.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17
Mean MD Anderson Symptom Inventory Scores at Baseline [Mean (Standard Deviation); unit: Scores on a scale] — The MD Anderson Symptoms Inventory (MDSAI) questionnaire evaluates 13 symptoms commonly experienced by patients with cancer with 6 additional items assessing the extent to which symptoms interfered with how patients feel and function. Scale is 0 (none), 1-4 (mild), 5-6 (moderate), and 7-10 (severe). A component score representing symptom severity is obtained by averaging the 13 symptom items (e.g., pain, fatigue, etc.) together. A component score representing symptom distress is obtaining by averaging the 6 symptom interference items (e.g., general activity, mood, etc.).
  Scores on a scale
    Symptom Severity Score | 2.0 (1.39)
    Symptom Interference Score | 2.94 (2.50)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Complete Response (CR) + Partial Response (PR)
Description: Complete Response + Partial Response was determined by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progressions. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 20 months
Measure: Count of Participants; unit: Participants
Arm/Group | PF-03084014 in Desmoid Tumors/Aggressive Fibromatosis
Number analyzed (Participants) | 17
Participants
  Complete Response | 0
  Partial Response | 5
  Not Evaluable | 1
  Stable Disease | 11
  Progressive Disease | 0

2. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 66 months and 27 days.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-03084014 in Desmoid Tumors/Aggressive Fibromatosis
Number analyzed (Participants) | 17
Participants | 17

3. Secondary Outcome: Number of Participants With Somatic or Germline Mutations Identified in Adenomatous Polyposis Coli Gene (APC) or Catenin Beta-1 (CTNNB1) Genes
Description: Tumor and blood samples were obtained from participants and genotyped for somatic and germline mutations.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | PF-03084014 in Desmoid Tumors/Aggressive Fibromatosis
Number analyzed (Participants) | 17
Participants | 15

4. Secondary Outcome: Mean MD Anderson Symptom Inventory Scores After Treatment
Description: The MD Anderson Symptoms Inventory (MDSAI) questionnaire includes questions regarding 13 symptoms commonly experienced by patients with cancer and 6 additional items that assess the extent to which these symptoms interfered with how patients felt and were able to function. The 0-10 scale (0=none, 1-4=mild, 5-6=moderate, and 7-10=severe) assesses how patients felt and were able to function over the previous 24 hours. A component score representing symptom severity is obtained by taking the average of the 13 symptom items (e.g., pain, fatigue, etc.) together. A component score representing symptom distress is obtaining by averaging the 6 symptom interference items (e.g., general activity, mood, etc.).
Time Frame: At baseline prior to drug administration and at least every 6 cycles of drug (18 weeks) up to 20 months of treatment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PF-03084014 in Desmoid Tumors/Aggressive Fibromatosis
Number analyzed (Participants) | 17
Scores on a scale
  Symptom Severity Score | 1.37 (1.46)
  Symptom Interference Score | 1.57 (2.69)

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 66 months and 27 days.
Arm/Group | PF-03084014 in Desmoid Tumors/Aggressive Fibromatosis
All-Cause Mortality (participants affected / at risk) | 1/17
Serious Adverse Events (participants affected / at risk) | 9/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-03084014 in Desmoid Tumors/Aggressive Fibromatosis (N=17)
Allergic reaction (Immune system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) — injury complications - Other, head contusion
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Surgical and medical procedures - Other, hysterectomy (Surgical and medical procedures) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-03084014 in Desmoid Tumors/Aggressive Fibromatosis (N=17)
Abdominal pain (Gastrointestinal disorders) | 8 (11)
Activated partial thromboplastin time prolonged (Investigations) | 4 (6)
Alanine aminotransferase increased (Investigations) | 9 (35)
Alkaline phosphatase increased (Investigations) | 5 (16)
Allergic rhinitis (Immune system disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 9 (23)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 12 (32)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (11)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (18)
Blood gonadotrophin abnormal (Investigations) | 1 (1)
Blurred vision (Eye disorders) | 3 (3)
Bronchial infection (Infections and infestations) | 1 (5)
Bruising (Injury, poisoning and procedural complications) | 5 (7)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac disorders - Other, potential murmur/"whooshing" (Cardiac disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 4 (5)
Cholesterol high (Investigations) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 2 (2)
Concentration impairment (Nervous system disorders) | 1 (2)
Confusion (Psychiatric disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Creatinine increased (Investigations) | 3 (13)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Depression (Psychiatric disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 15 (39)
Dizziness (Nervous system disorders) | 4 (8)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 7 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (5)
Dysgeusia (Nervous system disorders) | 3 (3)
Dysmenorrhea (Reproductive system and breast disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Ear and labyrinth disorders - Other, eustachian tube dysfunction (Ear and labyrinth disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Edema limbs (General disorders) | 6 (15)
Edema trunk (General disorders) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (2)
Endocrine disorders - Other, elevated glucose level (Endocrine disorders) | 1 (1)
Enterocolitis (Infections and infestations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Eye disorders - Other, eye injury (Eye disorders) | 1 (1)
Eye disorders - Other, left eye swelling & discharge (Eye disorders) | 1 (1)
Eye disorders - Other, macular degeneration - left eye (Eye disorders) | 1 (1)
Eye disorders - Other, vision changes (Eye disorders) | 1 (1)
Eye disorders - Other, visual disturbance (Eye disorders) | 1 (1)
Eye disorders - Other, exopthalmos bilateral (Eye disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 9 (14)
Fever (General disorders) | 6 (13)
Flatulence (Gastrointestinal disorders) | 2 (4)
Floaters (Eye disorders) | 1 (1)
Flu like symptoms (General disorders) | 6 (7)
Fracture (Injury, poisoning and procedural complications) | 4 (6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other, abdominal cramping (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, canker sores (Gastrointestinal disorders) | 1 (2)
Gastrointestinal disorders - Other, gastroenteritis (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (2)
Headache (Nervous system disorders) | 13 (22)
Hematoma (Vascular disorders) | 1 (1)
Hemoglobin increased (Investigations) | 1 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 8 (8)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (6)
Hypernatremia (Metabolism and nutrition disorders) | 2 (6)
Hypertension (Vascular disorders) | 7 (28)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (21)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 9 (14)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 8 (17)
Hypophosphatemia (Metabolism and nutrition disorders) | 13 (46)
Infections and infestations - Other, fungal infection (ear) (Infections and infestations) | 1 (1)
Infections and infestations - Other, oral infections (Infections and infestations) | 1 (1)
Infections and infestations - Other, rhinitis infective (Infections and infestations) | 1 (1)
Infections and infestations - Other, sinus infection (Infections and infestations) | 1 (3)
Infections and infestations - Other, upper respiratory infection (Infections and infestations) | 3 (3)
Infections and infestations - Other, viral gastroenteritis (Infections and infestations) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Injury, poisoning and procedural complications - Other, injury, abdomen contusion (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning and procedural complications - Other, injury, swollen mouth (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Investigations - Other, hypophosphatemia (Investigations) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 4 (4)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Libido decreased (Psychiatric disorders) | 3 (3)
Lip infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (2)
Lymphocyte count decreased (Investigations) | 12 (34)
Lymphocyte count increased (Investigations) | 1 (1)
Malaise (General disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 4 (5)
Menorrhagia (Reproductive system and breast disorders) | 3 (3)
Metabolism and nutrition disorders - Other, hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 6 (8)
Musculoskeletal and connective tissue disorder - Other, bone spur (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, right deltoid muscle tenderness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, stress injury (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, tendinitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, tendinitis left groin/thigh (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (10)
Nail infection (Infections and infestations) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 13 (27)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, cyst - right arm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Neoplasms benign, malignant and unspecified (incl cysts and polyps)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, popliteal cysts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, R paraspinal form tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — (incl cysts and polyps) - Other, sebaceous cyst (on back)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, rt groin area (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Nervous system disorders - Other, lightheadedness (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (8)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain (General disorders) | 8 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (9)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (5)
Paresthesia (Nervous system disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5)
Pharyngitis (Infections and infestations) | 2 (3)
Platelet count decreased (Investigations) | 4 (11)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Psychiatric disorders - Other, Mood swings (Psychiatric disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 7 (9)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (19)
Renal and urinary disorders - Other, elevated BUN (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, kidney stones (Renal and urinary disorders) | 1 (1)
Reproductive system and breast disorders - Other, amenorrhea (Reproductive system and breast disorders) | 3 (3)
Reproductive system and breast disorders - Other, breast tenderness (Reproductive system and breast disorders) | 1 (2)
Reproductive system and breast disorders - Other, elevated FSH (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast disorders - Other, elevated LH (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast disorders - Other, genital infection (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast disorders - Other, menstrual spotting (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast disorders - Other, menstruation (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast disorders - Other, R breat lump (Reproductive system and breast disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, cold (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, dry nasal passages (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Skin and subcutaneous tissue disorders - Other, cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, folliculitis (Skin and subcutaneous tissue disorders) | 4 (4)
Skin and subcutaneous tissue disorders - Other, skin keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, skin lesions (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, small hard lump/Rt upper thigh (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, left groin cystic lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, subcutaneous cysts (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin infection (Infections and infestations) | 7 (17)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Soft tissue necrosis upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Surgical and medical procedures - Other, esophageal dilation (Surgical and medical procedures) | 1 (1)
Surgical and medical procedures - Other, splenectomy (Surgical and medical procedures) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vaginal infection (Infections and infestations) | 2 (3)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (8)
Watering eyes (Ear and labyrinth disorders) | 1 (1)
Weight gain (Investigations) | 2 (14)
Weight loss (Investigations) | 4 (11)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 7 (17)
Wound infection (Infections and infestations) | 1 (1)
Psychiatric disorders - Other, Dreams (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT01981551/Prot_SAP_004.pdf
  • Informed Consent Form (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT01981551/ICF_005.pdf